CLINICAL TRIAL: NCT01611415
Title: A Clinical Pharmacological Study to Assess Pharmacodynamic and Pharmacokinetic Interactions Between Furosemide and Ipragliflozin in Healthy Subjects
Brief Title: Drug to Drug Interaction Study With Ipragliflozin and Furosemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1941-CL-0054; 2010-024071-98 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects; Pharmacokinetics of Ipragliflozin
Keywords: Phase 1; Ipragliflozin; Furosemide; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — ipragliflozin; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ipragliflozin (Experimental)
  Interventions: Drug: Ipragliflozin
- furosemide (Experimental)
  Interventions: Drug: Furosemide
- ipragliflozin & furosemide (Experimental)
  Interventions: Drug: Ipragliflozin; Drug: Furosemide

INTERVENTIONS:
Drug: Ipragliflozin — Oral
  Other Names: ASP1941
  Arms: ipragliflozin; ipragliflozin & furosemide
Drug: Furosemide — Oral
  Arms: furosemide; ipragliflozin & furosemide

SUMMARY:
A study to investigate if there are any pharmacodynamic and pharmacokinetic interactions between furosemide and ipragliflozin (ASP1941) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) more than or equal to 18.5 and less than 30.0 kg/m2

Exclusion Criteria:

* Any of the liver function tests above the upper limit of normal
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically)
* A QTc interval of >430 ms (males) or > 450 ms (females) consistently after duplicate measurements, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Assessment of urine sodium excretion, following multiple doses of furosemide alone compared to furosemide + ipragliflozin in healthy subjects | 6 days

SECONDARY OUTCOMES:
Assessment of urine sodium excretion, following multiple doses of ipragliflozin alone compared to furosemide + ipragliflozin in healthy subjects | 6 days
Assessment of pharmacodynamic parameters (i.e. calcium, chloride, potassium, phosphate and magnesium in blood and urine) following multiple doses of furosemide alone, ipragliflozin alone, and furosemide + ipragliflozin in healthy subjects | 9 days
Assessment of the pharmacokinetics of ipragliflozin when co-administered with furosemide compared to ipragliflozin alone | 10 days
  AUCtau (AUC during the time interval between consecutive dosing), Cmax (Maximum plasma concentration), t1/2 (Apparent Terminal Elimination Half-life) and tmax (Time to Attain Cmax)
Assessment of the pharmacokinetics of furosemide when co-administered with ipragliflozin compared to furosemide alone | 10 days
  AUCtau (AUC during the time interval between consecutive dosing), Cmax (Maximum plasma concentration), t1/2 (Apparent Terminal Elimination Half-life) and tmax (Time to Attain Cmax)
Assessment of the safety and tolerability of furosemide and ipragliflozin following multiple doses of furosemide alone, ipragliflozin alone, and furosemide + ipragliflozin in healthy subjects | 39 days
  Assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) and signs and symptoms of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Leeds, United Kingdom